CLINICAL TRIAL: NCT01119729
Title: Cardiovascular Diseases in HIV-infected Subjects (HIV-HEART Study)
Status: Completed | Type: Observational
Sponsor: University Hospital, Essen (Other)
Collaborators: Federal Ministry of Education and Reserach (BMBF) (Unknown)
Responsible Party: PD Dr. med. Till Neumann, FESC, Competence Network of Heart Failure
Other Study IDs: FKZ 01GI0205
Record Dates: First submitted 2010-05-07; First posted 2010-05-10 (Estimated); Last update posted 2010-05-10 (Estimated); Status verified 2010-05

CONDITIONS: Detection of Frequency, Severity and Progression of Cardiovascular Diseases in Patients With HIV-infection.; Effect on Cardiovascular Risk and Life Quality by Age, Gender, Classic Cardiovascular Risk Factors,; HIV-specific Cardiovascular Risk Factors, Cardiovascular Medication, Antiretroviral Medication
Keywords: Cardiac Diseases • HIV-Infection • AIDS • Antiretroviral Therapy
MeSH Terms: conditions — Coitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- HIV-infected Outpatients

SUMMARY:
Human immunodeficiency virus (HIV) infection has been associated with a variety of cardiovascular diseases. Even most industrialised countries exhibit a growing and aging population of HIV-infected patients in the majority treated with antiretroviral drugs, the investigators still do not know much about the impact of cardiovascular diseases in this group of patients. The present study is an ongoing trial that was conducted as a prospective and multicentre survey, being schemed to analyse the frequency and clinical course of cardiac disorders in HIV-infected patients.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Known HIV-infection
* Outpatients
* Written informed consent

Exclusion Criteria:

● Acute cardiovascular disease or unstable hemodynamic status in the three weeks before inclusion

• Pregnancy

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study population included outpatients who were at least 18 years of age, had a known HIV-infection and exhibited a stable disease status within 4 weeks before inclusion of the trial. Patients were recruited during a 20-month period in a consecutive manner from September 2004 to May 2006. Written informed consent was obtained from all participants
Sampling Method: Non-Probability Sample
Enrollment: 803 (Actual)

PRIMARY OUTCOMES:
Prevalence of cardiovascular diseases
  Prevalence of cardiovascular diseases including coronary artery disease, congestive heart failure, peripheral arterial disease, cerebrovascular events, and valvular diseases.

SECONDARY OUTCOMES:
Prevalence of cardiovascular disorders
  Prevalence of cardiovascular disorders determined by electrocardiography, exercise testing, echocardiography, blood samples.

CONTACTS AND LOCATIONS:
Locations (7):
- Germany (7):
  - Department of Dermatology, University Hospital of Bochum, Bochum, North Rhine-Westphalia
  - HIV Outpatient Department, Dortmund, North Rhine-Westphalia
  - HIV Outpatients Department, Duisburg, North Rhine-Westphalia
  - HIV Outpatient Department, Duisburg, North Rhine-Westphalia
  - Department of Dermatology, University Hospital of Essen, Essen, North Rhine-Westphalia
  - West German Heart Center Essen, Essen, North Rhine-Westphalia
  - HIV Outpatient Department, Essen, North Rhine-Westphalia

REFERENCES:
- [Background] Neumann T, Esser S, Potthoff A, Pankuweit S, Neumann A, Breuckmann F, Neuhaus K, Kondratieva J, Buck T, Muller-Tasch T, Wachter R, Prettin C, Gelbrich G, Herzog W, Pieske B, Rauchhaus M, Loffler M, Maisch B, Mugge A, Wasem J, Gerken G, Brockmeyer NH, Erbel R; HIV-HEART Study Investigative Group. Prevalence and natural history of heart failure in outpatient HIV-infected subjects: rationale and design of the HIV-HEART study. Eur J Med Res. 2007 Jun 27;12(6):243-8. PMID 17666313
- [Result] Neumann T. [HIV, AIDS and the cardiovascular risk]. Internist (Berl). 2008 Apr;49(4):429-30, 432-5. doi: 10.1007/s00108-008-2049-4. German. PMID 18305915
- [Result] Reinsch N, Buhr C, Krings P, Kaelsch H, Kahlert P, Konorza T, Neumann T, Erbel R; Competence Network of Heart Failure. Effect of gender and highly active antiretroviral therapy on HIV-related pulmonary arterial hypertension: results of the HIV-HEART Study. HIV Med. 2008 Aug;9(7):550-6. doi: 10.1111/j.1468-1293.2008.00602.x. Epub 2008 Jun 28. PMID 18557952
- [Result] Reinsch N, Buhr C, Krings P, Kaelsch H, Neuhaus K, Wieneke H, Erbel R, Neumann T; German Heart Failure Network. Prevalence and risk factors of prolonged QTc interval in HIV-infected patients: results of the HIV-HEART study. HIV Clin Trials. 2009 Jul-Aug;10(4):261-8. doi: 10.1310/hct1004-261. PMID 19723613
- [Result] Neumann T, Reinsch N, Neuhaus K, Brockmeyer N, Potthoff A, Esser S, Hower M, Neumann A, Mostardt S, Gelbrich G, Erbel R; fur die HIV-HEART-Studie sowie die Kompetenznetze Herzinsuffizienz und HIV/AIDS. [BNP in HIV-infected patients]. Herz. 2009 Dec;34(8):634-40. doi: 10.1007/s00059-009-3313-7. German. PMID 20024643
- [Derived] Reinsch N, Esser S, Gelbrich G, Brockmeyer N, Potthoff A, Schadendorf D, Erbel R, Neumann T. Valvular manifestations of human immunodeficiency virus infection--results from the prospective, multicenter HIV-HEART study. J Cardiovasc Med (Hagerstown). 2013 Oct;14(10):733-9. doi: 10.2459/JCM.0b013e32835dc953. PMID 24335884
- [Derived] Esser S, Gelbrich G, Brockmeyer N, Goehler A, Schadendorf D, Erbel R, Neumann T, Reinsch N. Prevalence of cardiovascular diseases in HIV-infected outpatients: results from a prospective, multicenter cohort study. Clin Res Cardiol. 2013 Mar;102(3):203-13. doi: 10.1007/s00392-012-0519-0. Epub 2012 Nov 2. PMID 23117698
- [Derived] Reinsch N, Kahlert P, Esser S, Sundermeyer A, Neuhaus K, Brockmeyer N, Potthoff A, Erbel R, Buck T, Neumann T. Echocardiographic findings and abnormalities in HIV-infected patients: results from a large, prospective, multicenter HIV-heart study. Am J Cardiovasc Dis. 2011;1(2):176-84. Epub 2011 Jul 30. PMID 22254197